CLINICAL TRIAL: NCT00651508
Title: Open Label, Multi-center, Phase 2 Study of KOS-1584 in Patients With Advanced or Metastatic Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) Previously Treated With First-Line Chemotherapy
Brief Title: Study to Evaluate KOS-1584 in Patients With Advanced or Metastatic Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA202-002; KOS-1584-203
Expanded Access: Available
Record Dates: First submitted 2008-03-26; First posted 2008-04-02 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Patients with Advanced or Metastatic stage IIIB/IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — KOS-1584

ARMS (1):
- Single Arm 25mg/m2 (Experimental): KOS-1584 25mg/m2
  Interventions: Drug: KOS-1584

INTERVENTIONS:
Drug: KOS-1584 — 25 mg/m2, IV (in the vein) on day 1 and 8 of each 21 day cycle until progression or unacceptable toxicity develops.
  Other Names: BMS-878271

SUMMARY:
The purpose of this study is to determine the Objective Response Rate of KOS-1584, as a single agent in patients with stage IIIB/IV NSCLC whose disease has progressed following initial chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven NSCLC, Stage IIIB or Stage IV.
* Eligible patients must have received only one prior chemotherapy regime for Stage IIIB/IV NSCLC.
* Good performance status.

Exclusion Criteria:

* Prior treatment with an epothilone.
* Known central nervous system (CNS) metastases.
* Any chemotherapy, radiation therapy or immunotherapy or any investigational agent (therapeutic or diagnostic) within 3 weeks prior to first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate of KOS-1584 | up to one year

SECONDARY OUTCOMES:
Progression Free Survival (PFS), Time to Progression (TTP), Time to Treatment Failure (TTF), time to response, duration of response, overall survival and safety of KOS-1584. | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Consultants In Blood Disorders & Cancer, Louisville, Kentucky, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx